CLINICAL TRIAL: NCT04348188
Title: Study of the Effectiveness of Supervised vs. Non-Supervised Therapeutic Exercise in Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Hospital Universitario Infanta Leonor (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20/007-E_TFM
Record Dates: First submitted 2020-02-28; First posted 2020-04-16 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer; Colon Cancer
Keywords: Quality of life; Terapeutic exercise; Cancer
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised exercise group (Experimental): Supervised intervention group: 3 weekly sessions of 1 hour during 6 weeks of therapeutic exercise in which aerobic physical activity will be combined with exercise strength of different muscle groups plus stretches on a supervised basis and strengthening of self-care.
  Interventions: Behavioral: Education program on healthy habits
- Not supervised exercise group (Active Comparator): Unsupervised intervention group: The same therapeutic exercise protocol will be scheduled which will be carried out autonomously without supervision with telephone tracking.
  Interventions: Behavioral: Education program on healthy habits

INTERVENTIONS:
Behavioral: Education program on healthy habits — 6-week supervised educational program with 12-month follow-up compared to the same unsupervised intervention

SUMMARY:
AIM:To evaluate the effectiveness of a therapeutic exercise program (PET) in cancer patients in improving the quality of life and the need for supervision by health professionals during the performance of same after 6 weeks of intervention. DESIGN: Randomized and controlled clinical trial, parallel groups with active control group. With masking of randomization, patient evaluation and analysis of the data. SUBJETS OF STUDY: 58 patients diagnosed with breast and colon cancer and treated up to 2 years later, both with surgery, chemotherapy and hormonal treatments (inhibitors of aromatase, tamoxifen). INTERVENTION: both groups the treatment will be a common work-based therapeutic exercise program aerobic, strength-resistance and self-stretching, in addition to a reinforcement in recommendations usual self-care. The study includes two phases, phase of supervised work and phase of tracing. One of the groups will be supervised in the realization of PET for a period of 6weeks and the other group will do it autonomously and without supervision. The patients will be followed for 1 year, with five blind evaluations: at the beginning of the study, after 6 weeks of intervention, 3, 6 and 12 months after the start of the study.MEASUREMENTS: Principal: Quality of life assessed with the questionnaire measured with the European questionnaire Organization for Research and Treatment of Cancer Quality of Life Questionnaire C-30 (EORTC QLQ-30). Pre-post intervention measure, 3, 6 and 12 months. Secondary: Cancer-related fatigue evaluated with the Functional Assessment of scale Chronic Illness Therapy - Fatigue (FACIT-F). Pre-post Measurement intervention, 3, 6 and 12 months. Functional capacity measured with the Test 6 minutes walking test. Pre-post Measurement intervention, 3, 6 and 12 months. Valuation of the measured force with manual hydraulic dynamometer and 5- test repetition sit-to-stand. Pre-post intervention measure, 3, 6 and 12 months.COST: effectiveness and cost / incremental utility associated to the program wil be estimated.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-70 years.
* Oncological stage I, II or III.
* Completed adjuvant treatment between 3 months to 2 years. ECOG 1-2.
* Sign informed consent

Exclusion Criteria:

* Inability to read, understand and complete questionnaires, read and understand a brochure explanatory, understand and follow verbal orders (example; illiteracy, dementia or blindness).
* Musculoskeletal disorders that prevent the exercise of the exercise bike, elliptical, march tape.
* Important neurological disorders that involve impaired balance, coordination, ataxia.
* Sporting activity at moderate intensity exceeding 150mnts / week.
* Symptomatic anemia.
* Fecal incontinence
* Patient with a digestive ostomy.
* Decompensated heart disease,
* Uncontrolled hypertension
* Heart failure.
* Musculoskeletal pathology (except for upper limb pathology in cancer patients of mom)
* Cardio-respiratory pathology that limits physical activity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Changes in Health Related Quality of Life: EORTC QLQ-30 | Basal, 1.5, 3, 6, 12 months follow up
  Quality of life assessed with the questionnaire measured with the European questionnaire Organization for Research and Treatment of Cancer Quality of Life Questionnaire C-30.
  (EORTC QLQ-30). The QLQ-C30 questionnaire is a specific questionnaire for cancer, it is composed of 30 questions or items that assess the quality of life in relation to physical, emotional, social aspects and in general the level of functionality of patients diagnosed with cancer. The QLQ-C30 questionnaire is assigned values between 1 and 4 (1: not at all, 2: a little, 3: a lot, 4: a lot) according to the patient's responses to the item, only in items 29 and 30 are assessed with score from 1 to 7 (1: bad, 7: excellent). The scores obtained are standardized and a score between 0 and 100 is obtained, 0 being the worst possible and 100 the best.

SECONDARY OUTCOMES:
Fatigue | Basal, 1.5, 3, 6, 12 months follow up
  Fatigue measurement with FACIT-F (Functional Assessment of Chronic Illness Therapy-Fatigue) questionaire.
  The FACIT-F 13-item scale is designed on a 5-point Likert scale (0 = nothing; 1 = little; 2 = something; 3 = a lot; 4 = very much). The FACIT-F scale is designed so that a high score is good, the possible score is 0 to 52, 0 being the worst possible and 52 the best.
Funtional capacity | Basal, 1.5, 3, 6, 12 months follow up
  The 6-minute walk test consists of measuring the maximum distance that the patient is able to walk in 6 minutes, on a tour short in a hallway, simultaneously assessing heart rate, oxygen saturation and degree of dyspnea. Usually healthy people can walk between 400 and 700 meters in 6 minutes, depending on age, height and sex
Valuation of the measured force | Basal, 1.5, 3, 6, 12 months follow up
  Valuation of the measured force with manual hydraulic dynamometer and 5- test repetition sit-to-stand. The test assesses the act of sitting and standing for five repetitions as quickly as possible, in a chair without arms with a seat height of 43 cm. The participant crosses his arms over his chest and sits with his back against the vertical back of the chair. The performance of the test is based on its duration; Consequently, the shorter the time it takes for the patient to perform the test, the better it will be.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Infanta Leonor, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No